CLINICAL TRIAL: NCT06819774
Title: Efficacy and Safety of Cetirizine Hydrochloride Injection in the Treatment of Acute Urticaria: a Randomized, Double-blind, Positive Controlled, Multicenter Phase III Clinical Study
Brief Title: Phase III Clinical Study of Cetirizine Hydrochloride Injection in Treatment of Acute Urticaria
Acronym: Phase III
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NTP-XTLQ-I-Ⅲ
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Acute Urticaria
Keywords: Cetirizine hydrochloride injection; acute urticatia
MeSH Terms: interventions — Cetirizine; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): Cetirizine hydrochloride injection；diphenhydramine hydrochloride injection simulator
  Interventions: Drug: Cetirizine Hydrochloride Injection
- Arm 2 (Experimental): diphenhydramine hydrochloride injection ；Cetirizine hydrochloride injection simulant
  Interventions: Drug: Diphenhydramine Hydrochloride Injection

INTERVENTIONS:
Drug: Cetirizine Hydrochloride Injection — The subjects received a single dose of 1-2 ml of the injection of cetirizine hydrochloride (administered by intravenous push) and a 1 ml dose of the injection simulant of diphenhydramine hydrochloride (administered by deep intramuscular injection), both as a simulation of a single administration.
  Other Names: Simulant of Diphenhydramine Hydrochloride Injection
  Arms: Arm 1
Drug: Diphenhydramine Hydrochloride Injection — The subjects received 1 ml of the injection of Diphenhydramine Hydrochloride (for deep intramuscular injection) and 1 ml of the injection of Simulated Cetirizine Hydrochloride (administered by rapid intravenous injection over 1 to 2 minutes), each as a single dose.
  Other Names: Simulant of Cetirizine Hydrochloride Injection
  Arms: Arm 2

SUMMARY:
The objective of this study was to evaluate the efficacy and safety of cetirizine hydrochloride injection in the treatment of acute urticaria.The participants were randomized to receive cetirizine hydrochloride or diphenhydramine hydrochloride.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18 - 65 years old (inclusive of the threshold value), gender not limited;
2. Diagnosed with acute urticaria (the definition of acute urticaria: spontaneous wheals and/or angioedema attacks ≤ 6 weeks);
3. At screening，the severity score of pruritus of the patient was ≥ 1 point ;
4. At screening，the degree score of wheals/erythema of the patient assessed by the investigator was ≥ 1 point ;
5. Be willing and able to give informed consent.

Exclusion Criteria:

1. Patients in whom an antihistamine are contraindicated (such as those with angle-closure glaucoma, symptomatic benign prostatic hyperplasia, etc.);
2. Patients who used H1 antagonists (such as diphenhydramine, cetirizine, loratadine, fexofenadine, levocetirizine, desloratadine, etc.) within 2 hours before randomization;
3. Patients who used H2 antagonists (such as cimetidine, ranitidine, famotidine, roxatidine, etc.) within 2 hours before randomization;
4. Patients who used doxepin within 2 hours before randomization;
5. Patients who received steroid hormone treatment for acute allergic reactions within 4 hours before randomization;
6. Patients who used epinephrine within 20 minutes before randomization;
7. Patients who are known to be allergic to hydroxyzine, cetirizine, levocetirizine, diphenhydramine;
8. Pregnant or lactating women; or those who have a pregnancy plan or plan to donate sperm/eggs from the screening day to the end of medication within 1 month; or those who are unwilling to take one or more contraceptive measures from the screening day to the end of medication within 1 month;
9. Patients with urticarial drug eruption;
10. Patients with acute urticaria who have concurrent symptoms such as laryngeal edema, allergic asthma, anaphylactic shock during screening;
11. Patients with urticarial vasculitis, hereditary angioedema, antihistamine-resistant urticaria or skin diseases that interfere with the evaluation of treatment efficacy during screening;
12. Patients with a history of immunodeficiency;
13. Patients with other major medical conditions (such as blood diseases, cardiovascular and cerebrovascular diseases, liver diseases, kidney diseases, etc.) or mental disorders and judged by the investigator to be unsuitable to participate in this study;
14. Patients who are concurrently using P-glycoprotein inhibitors (such as cyclosporine, itraconazole, dronedarone, amiodarone, quinidine, verapamil, etc.) during screening;
15. Patients who participated in other clinical trials within 3 months before screening (excluding those who only participated in the screening of the clinical trial but did not use the trial drugs or devices);
16. Patients with acute urticaria accompanied by fever during screening;
17. Patients engaged in dangerous jobs such as driving, high-altitude work, mechanical operation, etc., and cannot stop within 48 hours after medication;
18. Other various situations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Scoring of the severity of pruritus | Two hours after the treatment was completed
  Scoring of the severity of pruritus

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No